CLINICAL TRIAL: NCT04084119
Title: The Effect of Hypopressive Abdominal Exercise Versus General Strengthening Exercise on Abdominopelvic and Lumbar Function in Postpartum Women
Brief Title: Effect of Hypopressive Exercise Versus General Strengthening in Postpartum Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Mercè Balasch i Bernat, PhD Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H1545907781766
Record Dates: First submitted 2019-05-25; First posted 2019-09-10 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Postpartum Women
Keywords: postpartum; inter-rectus distance; diastasis recti; Lumbar disability; urinary incontinence; pelvic floor; quality of life
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants don't know to which intervention group they belong to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hypopressive abdominal exercise (Experimental): Participants will perform an hypopressive abdominal exercise program consisting of 18 sessions (6 weeks), 3 times a week, 30 minutes each session.
  Interventions: Other: hypopressive abdominal exercise
- general strengthening exercise (Active Comparator): Participants will perform a general strengthening exercise program consisting of 18 sessions (6 weeks), 3 times a week, 30 minutes each session.
  Interventions: Other: general strengthening exercise

INTERVENTIONS:
Other: hypopressive abdominal exercise — Participants will perform an hypopressive abdominal exercise program consisting of 18 sessions (6 weeks), 3 times a week, 30 minutes each session.
  Arms: hypopressive abdominal exercise
Other: general strengthening exercise — Participants will perform a general strengthening exercise program consisting of 18 sessions (6 weeks), 3 times a week, 30 minutes each session.
  Arms: general strengthening exercise

SUMMARY:
The aim of this study is to compare the effect of a hypopressive abdominal exercise program versus a general strengthening exercise program on inter-recti distance, abdominal and lumbar muscle thickness, lumbopelvic and abdominal pain and function, pelvic floor dysfunction, and quality of life in postpartum women. To evaluate the effects of the interventions, the subjects will be assessed at pre-intervention, immediately post-intervention and at 3-months follow-up.

DETAILED DESCRIPTION:
The aim of this study is to compare the effect of a hypopressive abdominal exercise program versus a general strengthening exercise program on inter-recti distance, abdominal and lumbar muscle thickness, lumbopelvic and abdominal pain and function, pelvic floor dysfunction, and quality of life in postpartum women. To evaluate the effects of the hypopressive exercise, the subjects will be assessed at pre-intervention, immediately post-intervention and at 3-months follow-up.

It will consist of a randomized controlled trial study. The sample will consist of women in the early postpartum period (6-8 weeks after delivery). Subjects will be randomly allocated to two different exercise programs: hypopressive abdominal exercise program and general strengthening exercise program. Both interventions will have a total duration of 6 weeks (18 sessions), 3 times a week, 30 minutes each session.

To evaluate the effects of the interventions, the subjects will be assessed at pre-intervention (6th-8th week postpartum), immediately post-intervention (12th-14th week postpartum) and at 3-months follow-up (24th-26th week postpartum). Inter-recti distance, abdominal and lumbar muscle thickness, lumbopelvic and abdominal pain and function, pelvic floor dysfunction, and quality of life will be measured.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 18-45 years old
* in the 6th-8th week postpartum
* both vaginal or caesarean delivery
* both primiparous or multiparous women

Exclusion Criteria:

* previous abdominal or pelvic surgery
* reasons to suspect metabolic, neurological or neuromuscular disease
* multiple birth delivery

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Inter-recti distance | pre-intervention
  Inter-recti distance will be measured by ultrasonography at rest, during abdominal draw-in and abdominal curl-up, at 2 locations on the linea alba (2 cm above and below the umbilicus).
Inter-recti distance | immediately post-intervention
  Inter-recti distance will be measured by ultrasonography at rest, during abdominal draw-in and abdominal curl-up, at 2 locations on the linea alba (2 cm above and below the umbilicus).
Inter-recti distance | 3-months follow-up
  Inter-recti distance will be measured by ultrasonography at rest, during abdominal draw-in and abdominal curl-up, at 2 locations on the linea alba (2 cm above and below the umbilicus).
Abdominal and lumbar muscles thickness | pre-intervention
  Transversus abdominis, obliquus internus, obliquus externus and multifidus thickness at rest and during draw-in will be measured by ultrasonography.
Abdominal and lumbar muscles thickness | immediately post-intervention
  Transversus abdominis, obliquus internus, obliquus externus and multifidus thickness at rest and during draw-in will be measured by ultrasonography.
Abdominal and lumbar muscles thickness | 3-months follow-up
  Transversus abdominis, obliquus internus, obliquus externus and multifidus thickness at rest and during draw-in will be measured by ultrasonography.

SECONDARY OUTCOMES:
Lumbopelvic and abdominal pain | pre-intervention
  Lumbopelvic and abdominal pain reported by the patient will be measured using a 100-mm visual analogue scale (VAS, 0-100, 0=minimum score, 100=maximum score). Lower values represent a better outcome (less pain).
Lumbopelvic and abdominal pain | immediately post-intervention
  Lumbopelvic and abdominal pain reported by the patient will be measured using a 100-mm visual analogue scale (VAS, 0-100, 0=minimum score, 100=maximum score). Lower values represent a better outcome (less pain).
Lumbopelvic and abdominal pain | 3-months follow-up
  Lumbopelvic and abdominal pain reported by the patient will be measured using a 100-mm visual analogue scale (VAS, 0-100, 0=minimum score, 100=maximum score). Lower values represent a better outcome (less pain).
Lumbopelvic and abdominal muscles function | pre-intervention
  Lumbopelvic and abdominal muscles function will be tested with the supine bridge test, the prone bridge test and the lateral bridge test.
Lumbopelvic and abdominal muscles function | immediately post-intervention
  Lumbopelvic and abdominal muscles function will be tested with the supine bridge test, the prone bridge test and the lateral bridge test.
Lumbopelvic and abdominal muscles function | 3-months follow-up
  Lumbopelvic and abdominal muscles function will be tested with the supine bridge test, the prone bridge test and the lateral bridge test.
Lumbar disability | pre-intervention
  Lumbar disability will be evaluated by the Oswestry Disability Index (ODI)
Lumbar disability | immediately post-intervention
  Lumbar disability will be evaluated by the Oswestry Disability Index (ODI)
Lumbar disability | 3-months follow-up
  Lumbar disability will be evaluated by the Oswestry Disability Index (ODI)
Severity of the urinary incontinence | pre-intervention
  The severity of the urinary incontinence will be assessed using the Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-IU-SF) (0-21).
Severity of the urinary incontinence | immediately post-intervention
  The severity of the urinary incontinence will be assessed using the Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-IU-SF) (0-21).
Severity of the urinary incontinence | 3-months follow-up
  The severity of the urinary incontinence will be assessed using the Incontinence Questionnaire-Urinary Incontinence Short Form (ICIQ-IU-SF) (0-21).
Sexual dysfunction | pre-intervention
  Sexual dysfunction will be assessed using the 6-item Female Sexual Function Index (FSFI-6) (5-30).
Sexual dysfunction | immediately post-intervention
  Sexual dysfunction will be assessed using the 6-item Female Sexual Function Index (FSFI-6) (5-30).
Sexual dysfunction | 3-months follow-up
  Sexual dysfunction will be assessed using the 6-item Female Sexual Function Index (FSFI-6) (5-30).
Self-reported quality of life | pre-intervention
  Self-reported quality of life will be evaluated with the Short Form-36 Health Survey (SF-36). In this scale, higher scores indicate higher quality of life.
Self-reported quality of life | immediately post-intervention
  Self-reported quality of life will be evaluated with the Short Form-36 Health Survey (SF-36). In this scale, higher scores indicate higher quality of life.
Self-reported quality of life | 3-months follow-up
  Self-reported quality of life will be evaluated with the Short Form-36 Health Survey (SF-36). In this scale, higher scores indicate higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Mercè B Balasch i Bernat, PhD, PT, Principal Investigator — Department of Physiotherapy. Faculty of Physioltherapy. Universitat de València
Locations (1):
- Mercè Balasch i Bernat, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No